CLINICAL TRIAL: NCT06159465
Title: Consensus Statements on the Utility of Defining ARDS and the Utility of Past and Current Definitions of ARDS--Protocol for a Delphi Study
Brief Title: Utility of Defining ARDS and Past and Current Definitions of ARDS
Acronym: Delphi_ARDS
Status: Completed | Type: Observational
Sponsor: NMC Specialty Hospital (Other)
Responsible Party: Principal Investigator, Prashant Nasa, HOD, Critical Care Medicine, NMC Specialty Hospital
Other Study IDs: ARDS_Delphi
Record Dates: First submitted 2023-11-25; First posted 2023-12-06 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Respiratory Distress Syndrome, Adult; Hypoxemic Respiratory Failure; Respiratory Failure; Phenotypic Abnormality; Delphi Study
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS), marked by acute hypoxemia and bilateral pulmonary infiltrates, has undergone multiple definitions over the years. Challenges persist regarding the ARDS definitions, leading to various revisions. Through the Delphi study, the investigators aims to gather global opinions on the conceptual framework of ARDS, assess the utility of current and past definitions, and explore the role of subphenotyping. The diverse panel's collective expertise will contribute valuable insights for refining future ARDS definitions and enhancing clinical management.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS), characterized by acute hypoxemia and bilateral pulmonary infiltrates that are not attributable to heart failure, has seen multiple definitions over the years. The primary purpose of a formal ARDS definition is to identify a homogenous cohort among patients with acute hypoxemic respiratory failure (AHRF), facilitating research, therapeutic trials, and prognostic assessment.

The validity of the conceptual framework of ARDS, however, has been challenged and uncertainties exist regarding the utility of ARDS definitions. Amongst other reasons, the lack of consensus on the conceptual model and diagnostic criteria have led to numerous revisions of the definition of ARDS. Furthermore, categorizing ARDS to assess treatment effects has had limited success, and subphenotypes have been proposed in part to address this issue.

The Delphi methodology has been used to generate expert consensus on components of the ARDS definition. Consensus process through a Delphi minimizes individual or professional dominance and peer pressure bias through a careful selection of experts, anonymous voting and monitoring attrition rates during Delphi rounds. A rigorous Delphi would be useful to assess the utility of the conceptual model of ARDS, past and current definitions of ARDS, and the value of categorisation of ARDS by means of subphenotyping.

Through this Delphi study, the investigators intend to assess the challenges in the conceptual framework of ARDS, past and current ARDS definitions, ongoing efforts in ARDS categorization and will develop consensus statements for future research in the definition and subphenotyping of ARDS.

ELIGIBILITY:
Inclusion Criteria:

* At least 5 years of clinical experience as a staff member, with care for AHRF or ARDS patients or preclinical expertise (of more than 5 years) in AHRF or ARDS;
* At least 5 publications (original studies) as a leading or senior author or member of the steering committee of an observational study or a randomised controlled trial in AHRF or ARDS;

Exclusion Criteria:

* Not more than 25% of panellists from the previous or current definitions of ARDS (including the Berlin Definition of ARDS, the Kigali Modification of the Definition of ARDS, and the New Global Definition of ARDS)
* Not more than 70% of the panellists from each sex; and from each of high and low-middle-income countries

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A diverse panel of 35 to 40 Panellists from different professional disciplines, such as Internal Medicine, Intensive Care Medicine, Respiratory Medicine, Anaesthesiology, and Physiology, with experience in the field of ARDS.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-04-07 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Consensus on the conceptual framework of ARDS, | 3-4 months
  Diverse group of panelist across the globe based on pre-specified qualification criteria and will conduct iterative Delphi rounds to generate consensus on the conceptual framework of ARDS.
Consensus on the utility of current and past definitions, | 3-4 months
  Diverse group of panelist across the globe based on pre-specified qualification criteria and will conduct iterative Delphi rounds to generate consensus on the utility of current and past definitions of ARDS.
Consensus on the role of subphenotyping in ARDS | 3-4 months
  Diverse group of panelist across the globe based on pre-specified qualification criteria and will conduct iterative Delphi rounds to generate consensus on the role of subphenotyping in ARDS

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Nasa, MD EDIC, Principal Investigator — HOD, Critical Care Medicine
Locations (1):
- NMC Specialty Hospital, Al Nahda, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
Anonymised reports of the Delphi rounds will be shared with original publication.

REFERENCES:
- [Result] Sweeney RM, McAuley DF. Acute respiratory distress syndrome. Lancet. 2016 Nov 12;388(10058):2416-2430. doi: 10.1016/S0140-6736(16)00578-X. Epub 2016 Apr 28. PMID 27133972
- [Result] Ranieri VM, Rubenfeld G, Slutsky AS. Rethinking Acute Respiratory Distress Syndrome after COVID-19: If a "Better" Definition Is the Answer, What Is the Question? Am J Respir Crit Care Med. 2023 Feb 1;207(3):255-260. doi: 10.1164/rccm.202206-1048CP. PMID 36150099
- [Result] Esteban A, Fernandez-Segoviano P, Frutos-Vivar F, Aramburu JA, Najera L, Ferguson ND, Alia I, Gordo F, Rios F. Comparison of clinical criteria for the acute respiratory distress syndrome with autopsy findings. Ann Intern Med. 2004 Sep 21;141(6):440-5. doi: 10.7326/0003-4819-141-6-200409210-00009. PMID 15381517
- [Result] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Result] Bos LDJ, Ware LB. Acute respiratory distress syndrome: causes, pathophysiology, and phenotypes. Lancet. 2022 Oct 1;400(10358):1145-1156. doi: 10.1016/S0140-6736(22)01485-4. Epub 2022 Sep 4. PMID 36070787
- [Result] Ferguson ND, Davis AM, Slutsky AS, Stewart TE. Development of a clinical definition for acute respiratory distress syndrome using the Delphi technique. J Crit Care. 2005 Jun;20(2):147-54. doi: 10.1016/j.jcrc.2005.03.001. PMID 16139155
- [Result] Matthay MA, Arabi Y, Arroliga AC, Bernard G, Bersten AD, Brochard LJ, Calfee CS, Combes A, Daniel BM, Ferguson ND, Gong MN, Gotts JE, Herridge MS, Laffey JG, Liu KD, Machado FR, Martin TR, McAuley DF, Mercat A, Moss M, Mularski RA, Pesenti A, Qiu H, Ramakrishnan N, Ranieri VM, Riviello ED, Rubin E, Slutsky AS, Thompson BT, Twagirumugabe T, Ware LB, Wick KD. A New Global Definition of Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2024 Jan 1;209(1):37-47. doi: 10.1164/rccm.202303-0558WS. PMID 37487152
- [Result] Nasa P, Jain R, Juneja D. Delphi methodology in healthcare research: How to decide its appropriateness. World J Methodol. 2021 Jul 20;11(4):116-129. doi: 10.5662/wjm.v11.i4.116. eCollection 2021 Jul 20. PMID 34322364
- [Result] Riviello ED, Kiviri W, Twagirumugabe T, Mueller A, Banner-Goodspeed VM, Officer L, Novack V, Mutumwinka M, Talmor DS, Fowler RA. Hospital Incidence and Outcomes of the Acute Respiratory Distress Syndrome Using the Kigali Modification of the Berlin Definition. Am J Respir Crit Care Med. 2016 Jan 1;193(1):52-9. doi: 10.1164/rccm.201503-0584OC. PMID 26352116
- [Derived] Nasa P, Bos LD, Estenssoro E, van Haren FM, Serpa Neto A, Rocco PR, Slutsky AS, Schultz MJ. Consensus statements on the utility of defining ARDS and the utility of past and current definitions of ARDS-protocol for a Delphi study. BMJ Open. 2024 Apr 25;14(4):e082986. doi: 10.1136/bmjopen-2023-082986. PMID 38670604